CLINICAL TRIAL: NCT00333775
Title: A Randomised, Double Blind, Placebo Controlled, Multicentre Study to Evaluate the Efficacy and Safety of Bevacizumab in Combination With Docetaxel in Comparison With Docetaxel Plus Placebo, as First Line Treatment for Patients With HER2 Negative Metastatic and Locally Recurrent Breast Cancer.
Brief Title: A Study of Bevacizumab (Avastin) in Women With HER2 Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BO17708; 2005-003862-40 (EudraCT Number)
Record Dates: First submitted 2006-06-05; First posted 2006-06-06 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Docetaxel 100 mg/m^2 plus placebo (Experimental): Participants received docetaxel 100 mg/m^2 intravenously on Day 1 of each 3 week cycle for a maximum of 27 weeks (9 cycles). In addition, participants received placebo to bevacizumab intravenously on Day 1 of each 3 week cycle until disease progression, unacceptable toxicity, or participant withdrawal.
  Interventions: Drug: Docetaxel; Drug: Placebo to bevacizumab
- Docetaxel 100 mg/m^2 plus bevacizumab 7.5 mg/kg (Experimental): Participants received docetaxel 100 mg/m^2 intravenously on Day 1 of each 3 week cycle for a maximum of 27 weeks (9 cycles). In addition, participants received bevacizumab 7.5 mg/kg intravenously on Day 1 of each 3 week cycle until disease progression, unacceptable toxicity, or participant withdrawal.
  Interventions: Drug: Docetaxel; Drug: Bevacizumab
- Docetaxel 100 mg/m^2 plus bevacizumab 15.0 mg/kg (Experimental): Participants received docetaxel 100 mg/m^2 intravenously on Day 1 of each 3 week cycle for a maximum of 27 weeks (9 cycles). In addition, participants received bevacizumab 15.0 mg/kg intravenously on Day 1 of each 3 week cycle until disease progression, unacceptable toxicity, or participant withdrawal.
  Interventions: Drug: Docetaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel was supplied in 2 vials, 1 containing docetaxel and 1 containing a solvent, for intravenous infusion.
Drug: Placebo to bevacizumab — Placebo to bevacizumab was supplied as a sterile liquid for intravenous infusion in single-use vials.
  Arms: Docetaxel 100 mg/m^2 plus placebo
Drug: Bevacizumab — Bevacizumab was supplied as a sterile liquid for intravenous infusion in single-use vials.
  Other Names: Avastin
  Arms: Docetaxel 100 mg/m^2 plus bevacizumab 15.0 mg/kg; Docetaxel 100 mg/m^2 plus bevacizumab 7.5 mg/kg

SUMMARY:
This study will evaluate the efficacy and safety of 2 doses of Avastin in combination with docetaxel, versus docetaxel plus placebo, in patients with metastatic HER2 negative breast cancer who are candidates for taxane-based chemotherapy but who have not received prior chemotherapy for metastatic disease. The anticipated time on treatment is 1-2 years and the target sample size is 500+ individuals.

DETAILED DESCRIPTION:
Five participants randomized to the docetaxel 100 mg/m^2 plus placebo group actually received docetaxel 100 mg/m^2 plus bevacizumab 7.5 mg/kg and are included in the docetaxel 100 mg/m^2 plus bevacizumab 7.5 mg/kg group for the adverse event results. Sixteen participants randomized to the docetaxel 100 mg/m^2 plus placebo group actually received docetaxel 100 mg/m^2 plus bevacizumab 15.0 mg/kg and are included in the docetaxel 100 mg/m^2 plus bevacizumab 15.0 mg/kg group for the adverse event results.

ELIGIBILITY:
Inclusion criteria:

* Female patients ≥ 18 years of age.
* Human epidermal growth factor receptor 2 (HER2)-negative cancer of the breast with locally recurrent or metastatic disease, suitable for chemotherapy.
* No adjuvant chemotherapy within 6 months before randomization, and no taxane-based chemotherapy within 12 months before randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion criteria:

* Previous chemotherapy for metastatic or locally recurrent breast cancer.
* Radiotherapy for treatment of metastatic disease.
* Other primary tumors within last 5 years, except for controlled limited basal cell or squamous cancer of the skin, or cancer in situ of the cervix.
* Spinal cord compression or brain metastases.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization.
* Inadequate bone marrow, liver, or renal function.
* Uncontrolled hypertension.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (106):
- Australia (8):
  - Adelaide, New South Wales
  - Camperdown, New South Wales
  - Westmead, New South Wales
  - Auchenflower, Queensland
  - Box Hill, Victoria
  - Fitzroy, Victoria
  - Ringwood East, Victoria
  - Perth, Western Australia
- Austria (4):
  - Graz
  - Salzburg
  - Vienna
  - Vöcklabruck
- Belgium (2):
  - Brussels
  - Wilrijk
- Brazil (6):
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Florianópolis, Santa Catarina
  - Barretos, São Paulo
  - São Paulo, São Paulo
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Greater Sudbury, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Beijing, China
- France (8):
  - Besançon
  - Bordeaux
  - Caen
  - Clermont-Ferrand
  - Dijon
  - Lille
  - Montpellier
  - Villejuif
- Germany (16):
  - Ansbach
  - Berlin
  - Düsseldorf
  - Erlangen
  - Frankfurt
  - Frankfurt am Main
  - Halle
  - Hamburg
  - Heidelberg
  - Jena
  - Lemgo
  - München
  - Stuttgart
  - Trier
  - Tübingen
  - Ulm
- Italy (9):
  - Bologna, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Trieste, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Treviglio, Lombardy
  - Biella, Piedmont
  - Taormina, Sicily
  - Macerata, The Marches
- Lithuania (2):
  - Kaunas
  - Vilnius
- Mexico (6):
  - Mexicali
  - Mexico City
  - Mérida
  - Monterrey
  - Obregón
  - Puebla City
- Netherlands (2):
  - Sittard
  - Utrecht
- Panama City, Panama
- Poland (5):
  - Krakow
  - Olsztyn
  - Poznan
  - Warsaw
  - Wroclaw
- Portugal (2):
  - Coimbra
  - Lisbon
- Bucharest, Romania
- South Africa (2):
  - Pretoria
  - Sandton
- Seoul, South Korea
- Spain (4):
  - Barcelona, Barcelona
  - Jaén, Jaen
  - Madrid, Madrid
  - Málaga, Malaga
- Sweden (3):
  - Linköping
  - Lund
  - Umeå
- Chur, Switzerland
- Taiwan (2):
  - Kaohsiung City
  - Taipei
- Thailand (2):
  - Bangkok
  - Khon Kaen
- United Kingdom (9):
  - Bournemouth
  - Cambridge
  - Edinburgh
  - Leeds
  - London
  - Manchester
  - Middlesex
  - Newcastle upon Tyne
  - Truro

REFERENCES:
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants randomized to the placebo group received bevacizumab 7.5 mg/kg (n=5) or 15.0 mg/kg (n=16). Please see the Detailed Description for an explanation of the differences in the number of participants in the treatment groups in Participant Flow and Adverse Events.
Period: Overall Study
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg
Started | 241 | 248 | 247
Received Treatment | 238 | 247 | 245
Completed | 0 | 0 | 0
Not Completed | 241 | 248 | 247
Not completed — Death | 144 | 149 | 143
Not completed — In Follow-up When Study Stopped | 87 | 92 | 96
Not completed — Lost to Follow-up | 10 | 7 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants, regardless of whether they received study drug or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg | Total
Number analyzed (Participants) | 241 | 248 | 247 | 736
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (10.47) | 53.9 (10.61) | 53.6 (10.78) | 53.7 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 248 | 247 | 736
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was evaluated using Response Evaluation Criteria In Solid Tumors (RECIST 1.0). Progression-free survival was defined as the time from randomization to the time of the first documented disease progression or death, whichever occurred first. Disease progression was defined as ≥ 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the unequivocal progression of existing non-target lesions, or appearance of new lesion(s).
Time Frame: Baseline to the 15 Sep 2008 cut-off date (up to 2 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether they received study drug or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg
Number analyzed (Participants) | 241 | 248 | 247
Months | 8.0 [7.2 to 8.3] | 8.7 [8.2 to 9.9] | 8.8 [8.4 to 10.2]
Statistical Analysis 1: Comparison: Docetaxel 100 mg/m^2 Plus Placebo vs Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg; Test type: Superiority or Other; p = 0.0318, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.63 to 0.98]
Statistical Analysis 2: Comparison: Docetaxel 100 mg/m^2 Plus Placebo vs Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg; Test type: Superiority or Other; p = 0.0036, Log Rank; Hazard Ratio, log = 0.72, 95% CI 2-sided [0.57 to 0.90]

2. Secondary Outcome: Percentage of Participants With a Complete Response or a Partial Response
Description: Responses were evaluated using the Response Evaluation Criteria in Solid Tumors. A complete response was defined as the disappearance of all target lesions or the disappearance of all non-target lesions and normalization of tumor marker level. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Baseline to the 15 Sep 2008 cut-off date (up to 2 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether they received study drug or not. Only participants with measurable disease at Baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg
Number analyzed (Participants) | 207 | 201 | 206
Percentage of participants
  Complete response | 1.0 [0.1 to 3.4] | 3.0 [1.1 to 6.4] | 1.0 [0.1 to 3.5]
  Partial response | 43.5 [36.6 to 50.5] | 52.2 [45.1 to 59.3] | 62.1 [55.1 to 68.8]

3. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first documented complete response or partial response to disease progression or death. A complete response was defined as the disappearance of all target lesions or the disappearance of all non-target lesions and normalization of tumor marker level. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Responses were evaluated using the Response Evaluation Criteria in Solid Tumors.
Time Frame: Baseline to the 15 September 2008 cut-off date (up to 2 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether they received study drug or not. Only participants with measurable disease at Baseline who had a complete response or a partial response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg
Number analyzed (Participants) | 92 | 111 | 130
Months | 6.4 [5.8 to 6.9] | 7.2 [6.4 to 9.1] | 7.0 [6.4 to 8.5]

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as time from randomization to the date of disease progression, death, or withdrawal of treatment due to an adverse event, withdrawal of informed consent, insufficient therapeutic response, refusal of treatment/failure to co-operate, or failure to return, whichever occurred first.
Time Frame: Baseline to the 15 September 2008 cut-off date (up to 2 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether they received study drug or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg
Number analyzed (Participants) | 241 | 248 | 247
months | 6.1 [5.6 to 7.0] | 7.0 [6.1 to 7.7] | 7.7 [7.1 to 8.0]
Statistical Analysis 1: Comparison: Docetaxel 100 mg/m^2 Plus Placebo vs Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg; Test type: Superiority or Other; p = 0.1105, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.04]
Statistical Analysis 2: Comparison: Docetaxel 100 mg/m^2 Plus Placebo vs Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg; Test type: Superiority or Other; p = 0.0241, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.65 to 0.97]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to death from any cause.
Time Frame: Baseline to the 15 Sep 2008 cut-off date (up to 2 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether they received study drug or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg
Number analyzed (Participants) | 241 | 248 | 247
Months | NA [NA to NA] — Due to the low number of events, the median and lower and upper limits of the 95% confidence interval could not be reliably estimated. | NA [15.7 to NA] — Due to the low number of events, the median and upper limit of the 95% confidence interval could not be reliably estimated. | NA [14.9 to NA] — Due to the low number of events, the median and upper limit of the 95% confidence interval could not be reliably estimated.
Statistical Analysis 1: Comparison: Docetaxel 100 mg/m^2 Plus Placebo vs Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg; Test type: Superiority or Other; p = 0.6962, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.62 to 1.37]
Statistical Analysis 2: Comparison: Docetaxel 100 mg/m^2 Plus Placebo vs Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg; Test type: Superiority or Other; p = 0.0765, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.45 to 1.04]

ADVERSE EVENTS:
Description: Safety population: All randomized participants exposed to study medication.
  Please see the Detailed Description for an explanation of the differences in the number of participants in the treatment groups in Participant Flow and Adverse Events.
Arm/Group | Docetaxel 100 mg/m^2 Plus Placebo | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 82/217 | 106/252 | 120/261
Other Adverse Events (participants affected / at risk) | 216/217 | 251/252 | 260/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel 100 mg/m^2 Plus Placebo (N=217) | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg (N=252) | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg (N=261)
Febrile neutropenia (Blood and lymphatic system disorders) | 21 | 29 | 37
Neutropenia (Blood and lymphatic system disorders) | 4 | 13 | 18
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Infection (Infections and infestations) | 5 | 3 | 2
Neutropenic sepsis (Infections and infestations) | 2 | 3 | 2
Pneumonia (Infections and infestations) | 4 | 2 | 1
Neutropenic infection (Infections and infestations) | 2 | 2 | 1
Anal abscess (Infections and infestations) | 0 | 2 | 2
Central line infection (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 3 | 0
Sepsis (Infections and infestations) | 0 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 2 | 0
Anal infection (Infections and infestations) | 0 | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Catheter bacteraemia (Infections and infestations) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 1
Catheter sepsis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Lung abscess (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Nail bed infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Periodontal infection (Infections and infestations) | 0 | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Stent related infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 8
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 6 | 7
Asthenia (General disorders) | 1 | 6 | 4
Mucosal inflammation (General disorders) | 1 | 1 | 2
Oedema peripheral (General disorders) | 2 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0
General physical health deterioration (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 1 | 0
Catheter related complication (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 1
Ill-defined disorder (General disorders) | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Cranial nerve palsies multiple (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 0
Microangiopathy (Vascular disorders) | 2 | 0 | 0
Embolism venous (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Central venous catheter removal (Surgical and medical procedures) | 0 | 0 | 1
Vertebroplasty (Surgical and medical procedures) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel 100 mg/m^2 Plus Placebo (N=217) | Docetaxel 100 mg/m^2 Plus Bevacizumab 7.5 mg/kg (N=252) | Docetaxel 100 mg/m^2 Plus Bevacizumab 15.0 mg/kg (N=261)
Fatigue (General disorders) | 96 | 105 | 109
Asthenia (General disorders) | 83 | 88 | 97
Mucosal inflammation (General disorders) | 48 | 87 | 78
Oedema peripheral (General disorders) | 89 | 63 | 61
Pyrexia (General disorders) | 45 | 61 | 63
Oedema (General disorders) | 32 | 12 | 21
Pain (General disorders) | 20 | 16 | 16
Chest pain (General disorders) | 19 | 10 | 20
Malaise (General disorders) | 6 | 10 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 154 | 181 | 183
Nail disorder (Skin and subcutaneous tissue disorders) | 87 | 118 | 118
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 47 | 80 | 70
Rash (Skin and subcutaneous tissue disorders) | 43 | 43 | 47
Dry skin (Skin and subcutaneous tissue disorders) | 32 | 33 | 25
Erythema (Skin and subcutaneous tissue disorders) | 20 | 26 | 33
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 28 | 23
Onycholysis (Skin and subcutaneous tissue disorders) | 9 | 21 | 25
Skin exfoliation (Skin and subcutaneous tissue disorders) | 11 | 21 | 20
Nail toxicity (Skin and subcutaneous tissue disorders) | 15 | 16 | 12
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 | 14 | 10
Diarrhoea (Gastrointestinal disorders) | 106 | 143 | 140
Nausea (Gastrointestinal disorders) | 117 | 115 | 132
Stomatitis (Gastrointestinal disorders) | 60 | 127 | 115
Constipation (Gastrointestinal disorders) | 64 | 89 | 77
Vomiting (Gastrointestinal disorders) | 59 | 64 | 75
Abdominal pain (Gastrointestinal disorders) | 39 | 45 | 58
Dyspepsia (Gastrointestinal disorders) | 27 | 36 | 43
Abdominal pain upper (Gastrointestinal disorders) | 34 | 24 | 32
Haemorrhoids (Gastrointestinal disorders) | 14 | 22 | 22
Toothache (Gastrointestinal disorders) | 13 | 13 | 14
Dysphagia (Gastrointestinal disorders) | 12 | 13 | 13
Dry mouth (Gastrointestinal disorders) | 8 | 15 | 12
Gingivitis (Gastrointestinal disorders) | 4 | 11 | 16
Headache (Nervous system disorders) | 56 | 86 | 79
Dysgeusia (Nervous system disorders) | 59 | 77 | 63
Peripheral sensory neuropathy (Nervous system disorders) | 60 | 67 | 63
Paraesthesia (Nervous system disorders) | 40 | 46 | 51
Neuropathy peripheral (Nervous system disorders) | 30 | 35 | 26
Dizziness (Nervous system disorders) | 25 | 26 | 31
Hypoaesthesia (Nervous system disorders) | 11 | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 80 | 82 | 88
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 | 74 | 90
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 | 56 | 44
Back pain (Musculoskeletal and connective tissue disorders) | 45 | 36 | 44
Bone pain (Musculoskeletal and connective tissue disorders) | 38 | 35 | 42
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 | 34 | 36
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 14 | 17
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 | 12 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 16 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 47 | 123 | 128
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 67 | 61
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 | 44 | 60
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 | 26 | 38
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 27 | 28
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 24 | 28
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 | 10 | 17
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 13 | 12
Lacrimation increased (Eye disorders) | 63 | 114 | 120
Conjunctivitis (Eye disorders) | 11 | 16 | 39
Upper respiratory tract infection (Infections and infestations) | 23 | 22 | 28
Nasopharyngitis (Infections and infestations) | 14 | 20 | 35
Urinary tract infection (Infections and infestations) | 18 | 27 | 20
Influenza (Infections and infestations) | 12 | 26 | 15
Rhinitis (Infections and infestations) | 9 | 11 | 18
Sinusitis (Infections and infestations) | 8 | 10 | 19
Neutropenia (Blood and lymphatic system disorders) | 44 | 51 | 53
Anaemia (Blood and lymphatic system disorders) | 37 | 34 | 32
Leukopenia (Blood and lymphatic system disorders) | 14 | 21 | 20
Hypertension (Vascular disorders) | 32 | 44 | 66
Hot flush (Vascular disorders) | 16 | 16 | 19
Flushing (Vascular disorders) | 12 | 15 | 19
Lymphoedema (Vascular disorders) | 15 | 19 | 8
Decreased appetite (Metabolism and nutrition disorders) | 58 | 78 | 85
Insomnia (Psychiatric disorders) | 34 | 31 | 35
Depression (Psychiatric disorders) | 11 | 13 | 13
Anxiety (Psychiatric disorders) | 8 | 11 | 16
Weight decreased (Investigations) | 12 | 29 | 30
Weight increased (Investigations) | 16 | 5 | 7
Proteinuria (Renal and urinary disorders) | 8 | 12 | 24
Vertigo (Ear and labyrinth disorders) | 10 | 11 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.